CLINICAL TRIAL: NCT05257850
Title: Management of Breathlessness with High-flow Nasal Therapy or a Fan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Juho Lehto, MD,PhD,Professor, Tampere University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R20049
Record Dates: First submitted 2022-01-16; First posted 2022-02-25 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Breathlessness; Cancer
MeSH Terms: conditions — Dyspnea; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fan first (Active Comparator): Patients use the fan first and high-flow nasal therapy thereafter
  Interventions: Device: High-flow nasal therapy; Device: Airflow directed to face by a fan
- High-flow nasal therapy first (Active Comparator): Patients use high-flow nasal therapy first and the fan thereafter
  Interventions: Device: High-flow nasal therapy; Device: Airflow directed to face by a fan

INTERVENTIONS:
Device: High-flow nasal therapy — A high-flow nasal therapy for 30 minutes.
Device: Airflow directed to face by a fan — A fan directed to the face for 30 minutes

SUMMARY:
Airflow directed to the face by a fan is shown to relief breathlessness in palliative care and some studies have suggested High-Flow nasal airflow therapy beneficial as well. However, these two treatments have not been compared.

40 patients with advanced cancer and breathlessness are recruited from Tampere University Hospital or Pirkanmaa Hospice. All patients are treated with two therapies: 1. High-Flow nasal airflow therapy with a nasal cannula and 2. airflow directed to the face by a fan. Both treatment periods last 30 minutes or as long as the patient wish to use the therapy. The effects of the therapies on breathlessness are compared by asking the subjective relief of breathlessness after each therapies. The study do not limit any other therapies used in the normal clinical care for the patients. Thus, all the other therapies the physicians taking care of the patient orders are permitted. Hopefully, the patients achieve relief for their breathlessness through the study treatments given in addition to their normal treatment. There are no significant risks related to the therapies, but they may cause some inconveniences such as mouth dryness. These possible side-effects of the therapies are asked as well.

DETAILED DESCRIPTION:
Airflow directed to the face by a fan is shown to relief breathlessness in palliative care and some studies have suggested High-Flow nasal airflow therapy beneficial as well. However, these two treatments have not been compared and High-Flow nasal airflow therapy has not been tested in the context of hospice.

40 patients over 18 years with advanced cancer and breathlessness are recruited from Tampere University Hospital or Pirkanmaa Hospice. All patients are treated with two therapies: 1. High-Flow nasal airflow therapy with a nasal cannula and 2. airflow directed to the face by a fan (crossover trial). Both treatment periods last 30 minutes or as long as the patient wish to use the therapy. The effects of the therapies on breathlessness are compared by asking the subjective relief of breathlessness after each therapies with numeric rating scale (NRS) from 0 (no breathlessness) to 10 (the worst possible breathlessness). Influence of the treatments on anxiety, pain and mouth dryness are measured as well with numeric rating scale (NRS) from 0 to 10. The study do not limit any other therapies used in the normal clinical care for the patients. Thus, all the other therapies the physicians taking care of the patient orders are permitted. Hopefully, the patients achieve relief for their breathlessness through the study treatments given in addition to their normal treatment. There are no significant risks related to the therapies, but they may cause some inconveniences such as mouth dryness. These possible side-effects of the therapies are asked as well.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer
* At least 18 years of age
* Breathlessness (At least 3 on a NRS-scale from 0 to 10)
* Capable to understand the study and to give informed consent
* Do not benefit from ICU treatment or resuscitation defined by the physician taking care of the patient

Exclusion Criteria:

* Insufficient co-operation for the study treatment or to give informed consent
* Oxygen saturation under 88 % on room air
* Need for other device to treat the breathlessness
* The reason of breathlessness can be immediately treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Breathlessness after the study treatments (difference between the High-Flow Nasal Therapy and a fan) | Measurements are made immediately before and immediately after the treatment period.
  The breathlessness after the study treatments measured by numeric rating scale (NRS) from 0 (no breathlessness) to 10 (the worst possible breathlessness).

SECONDARY OUTCOMES:
Change in breathlessness before and after the treatments | Measurements are made immediately before and immediately after the treatment period.
  Change in breathlessness before and after the treatments measured by numeric rating scale (NRS) from 0 (no breathlessness) to 10 (the worst possible breathlessness).
Change in mouth dryness before and after the treatments | Measurements are made immediately before and immediately after the treatment period.
  Change in mouth dryness before and after the treatments measured by numeric rating scale (NRS) from 0 (no mouth dryness) to 10 (the worst possible mouth dryness).
Change in anxiety before and after the treatments | Measurements are made immediately before and immediately after the treatment period.
  Change in anxiety before and after the treatments measured by numeric rating scale (NRS) from 0 (no anxiety) to 10 (the worst possible anxiety).
Change in pain before and after the treatments | Measurements are made immediately before and immediately after the treatment period.
  Change in pain before and after the treatments measured by numeric rating scale (NRS) from 0 (no pain) to 10 (the worst possible pain).
Change in respiratory frequency with the treatments | Measurements are made immediately before and immediately after the treatment period.
  Change in respiratory frequency measured by calculating breaths per minute.
Change in heart rate with the treatments | Measurements are made immediately before and immediately after the treatment period.
  Change in heart rate measured by calculating heart beats per minute.
Change in oxygen saturation with the treatments | Measurements are made immediately before and immediately after the treatment period.
  Change in peripheral oxygen saturation (%) measured with pulse oximeter.
Proportion of patients reporting to have overall benefit of the treatments | Opinion is asked immediately after the treatment
  Proportion of patients reporting to have overall benefit of the treatments
Proportion of patients who report side-effects of the treatments | Experienced side-effects are asked immediately after the treatment
  Proportion of patients who report side-effects of the treatments

CONTACTS AND LOCATIONS:
Overall Officials: Juho Lehto, Professor, Principal Investigator — Tampere University Hospital
Locations (2):
- Finland (2):
  - Pirkanmaa Hospice, Tampere
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leivo-Korpela S, Rantala HA, Lehtimaki L, Piili RP, Hasala H, Korhonen T, Lehto JT. Management of Dyspnea With High-Flow Nasal Air or Fan-A Randomized Controlled Crossover Trial. J Pain Symptom Manage. 2026 Jan;71(1):8-15. doi: 10.1016/j.jpainsymman.2025.08.033. Epub 2025 Sep 4. PMID 40914402